CLINICAL TRIAL: NCT03968276
Title: Study of the Interest of Patients Undergoing Anti-thrombotic Treatment in a Digital Application of Therapeutic Assistance
Acronym: APPLIAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI decided to stop the study.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APPLIAC
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Vascular Diseases
Keywords: antithrombotic treatment; digital therapeutic application assistance
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- use of digital tablet (Experimental): if the patient is included in the study, an educational tablet (digital tablet) is given to the patient.
  The first connection to the tablet and then to the "My medication protects my vessels" application is made by the investigator in the presence of the patient. The application is configured by the investigator with the choice of the vascular pathology(s) corresponding to the patient included and the prescribed anti-thrombotic treatments. Thus, for each patient, the content of the tablet is adapted and personalized according to his vascular profile.
  After discharge from hospital, the patient has the educational tablet at his disposal for 1 month at home. The application offers patients various information supports (tools, questionnaires and pill box). Throughout its use, it may contact the investigating physician via a telephone number available within the application if it encounters a problem related to the study.
  Interventions: Other: use of digital tablet

INTERVENTIONS:
Other: use of digital tablet — At the end of hospitalization, the patient has an educational tablet at his disposal for 1 month at home. Throughout its use, the patient may contact the investigating physician via a telephone number available within the application if he/she encounters a problem related to the study. At the end of this month, the patient must complete two questionnaires through the application to assess his or her knowledge of his or her condition and treatment, as well as his or her satisfaction with the use of the tablet.
  In this research, 1 month after inclusion, the patient will have an additional follow-up visit corresponding to a dedicated consultation in the vascular medicine department. It will allow the patient to review the use of the tablet and his or her satisfaction with the use of such a tool.

SUMMARY:
Medical ethics encourages medical personal to actively care for patients, however old they may be, if they have maintained their physical autonomy and mental integrity to travel the path of medical care together. Many of the patients are in this situation today and their age does not seem to be a limiting factor in the care required.

For more than 60 years, antithrombotics have played a major role in the management of thromboembolic and arterioatheromatous diseases. the doctors have therefore seen the advent of low molecular weight heparins, new platelet antiaggregants and then direct oral anticoagulants.

If their contribution is no longer discussed today, it is necessary to take into consideration the risks they cause, particularly in terms of haemorrhage. Indeed, antithrombotics are the leading cause of serious adverse reactions in France with anti-vitamins K (AVK) which are the leading cause of hospitalization for severe iatrogeny in France. This risk is increased by the coexistence of haemorrhagic risk factors: drug interaction, misuse, failure to comply with contraindications and precautions for use, especially as exposure to these drugs increases with age.

DETAILED DESCRIPTION:
The risk of bleeding varies in different populations and according to the treatment used. Severe bleeding under AVK has an incidence of 0.6 to 10% per year. Fatal hemorrhage is in the order of 1%. The risk factors for bleeding are controversial: history of bleeding in the patient, instability of the International Normalized Ratio (INR) at the time of introduction of KVAs and during the first few months, poor patient compliance, drug combinations (antiplatelet, non-steroidal anti-inflammatory drugs: NSAIDs, paracetamol, etc.) or association with alcohol. National pharmacovigilance data indicate that serious accidents are not uncommon due to frequent misuse of antithrombotics in common practice.

There are risk factors related to the patient and his or her comorbidities: history of bleeding, stroke, comorbidities such as age > 65 years, diabetes, cancer, chronic renal failure.

Despite the various aids to therapeutic patient education (surveillance logbook, computerised INR monitoring), there has been no decrease in the frequency of iatrogenic accidents, either in hospitals or in urban medicine.

The use of smartphone applications in the medical field is increasingly evolving among healthcare professionals and patients. They allow for more personalized care, and can also promote interaction with health professionals.

Strengthening the link between specialist doctors and the general practitioner for joint patient management will improve their follow-up and reduce the risk of iatrogeny.

In 2016, a survey was conducted in the vascular medicine department of the Groupe Hospitalier Paris Saint-Joseph (GHPSJ) to assess access to smartphones among patients on anti-thrombotic medication. Of the 100 patients enrolled, 74 were on anticoagulant or platelet aggregation therapy. Of these, 50 had a mobile phone and 24% used the Internet and made downloads to their phones.

This raises the question of the interest that patients might have in a mobile application on the use of anti-thrombotics. As the profile of patients seen in hospital is different from those consulting in general medicine, it seems interesting to study these two populations in order to know if there is a difference in their attitude towards the smartphone.

In order to find a new way to limit the iatrogeny of antithrombotic drugs, the investigators wanted to set up a medical application (educational tablet) for patients to provide them with support to better manage their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient hospitalized in the vascular medicine department of the GHPSJ or attending a general medical consultation at the CMT
* Patient with at least one vascular pathology: pulmonary embolism, venous thrombosis or phlebitis, cardiac arrhythmia by atrial fibrillation, obliterating arteriopathy of the lower limbs or myocardial infarction
* Patient on antithrombotic treatment[anticoagulants : AVK or Anticoagulants Oraux Directs (AOD), or antiplatelet agents]
* Patient affiliated to a health insurance plan
* Patient able to read and understand the French language
* Patient capable of giving free, informed and express consent

Exclusion Criteria:

* Patient not residing in Ile de France
* Patient whose investigator considers that he/she is not able to use a digital tablet
* Patient deprived of liberty
* Patient under guardianship or curatorship
* Refusal to participate in the study
* Patient judged not to be included by the investigator on the basis of the inclusion questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Return of the tablet in working order and to its use | 1 month
  return (yes/no) and use

SECONDARY OUTCOMES:
Number of pages consulted on the educational tablet | 1 month
Analyses of patient treatment knowledge assessment questionnaires | Day 0 - 1 month
  The two questionnaires contain 12 and 11 questions respectively. the possible answers are yes or no
Analogical visual scale of patient satisfaction | 1 month
  Analogical visual scale of patient satisfaction from minimum 0 (very satisfied) to maximum 10 (not satisfied)
Questionnaire on compliance with antithrombotic treatments on application | 1 month
  taking antithrombotic treatments (yes/no)
Reporting of adverse events via the dedicated field on the educational tablet | 1 month
Number of calls from city physicians and pharmacists received by the investigator | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Parinaz GHAFFARI, MD, Study Director — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Linkins LA, Choi PT, Douketis JD. Clinical impact of bleeding in patients taking oral anticoagulant therapy for venous thromboembolism: a meta-analysis. Ann Intern Med. 2003 Dec 2;139(11):893-900. doi: 10.7326/0003-4819-139-11-200312020-00007. PMID 14644891
- [Result] Dahri K, Loewen P. The risk of bleeding with warfarin: a systematic review and performance analysis of clinical prediction rules. Thromb Haemost. 2007 Nov;98(5):980-7. PMID 18000602